CLINICAL TRIAL: NCT05601284
Title: Psychological Intervention for Misophonia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12981
Record Dates: First submitted 2022-10-26; First posted 2022-11-01 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2023-12

CONDITIONS: Misophonia
MeSH Terms: conditions — misophonia | interventions — Acceptance and Commitment Therapy; Autogenic Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and commitment therapy (Experimental): ACT teaches skills to develop acceptance, mindfulness, and defusion from difficult internal experiences while increasing connections with personal values and encouraging meaningful behavioral changes. ACT for misophonia combines core ACT processes with a traditional audiological behavioral intervention for a integrated, multi-disciplinary approach for the assessment and treatment of misophonia. Treatment begins with a brief focus on the behavioral intervention, followed by the teaching of ACT skills to support the use of the behavioral methods. The intervention consists of 12 total individual sessions of ACT+behavioral management.
  Interventions: Behavioral: Acceptance and commitment therapy
- Progressive relaxation training (Active Comparator): PRT for misophonia consists of basic psychoeducation for misophonia followed by PRT. PRT involves learning to tense and relax muscles. Early sessions focus on tensing and relaxing smaller muscle groups, while later sessions focus on larger muscle groups. Final sessions focus on relaxation as produced by recalling previous relaxation and a review of skills learned. PRT consists of 12 individual total sessions.
  Interventions: Behavioral: Progressive relaxation training

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy — ACT teaches skills to develop acceptance, mindfulness, and defusion from difficult internal experiences while increasing connections with personal values and encouraging meaningful behavioral changes. ACT for misophonia combines core ACT processes with a traditional audiological behavioral intervention for a integrated, multi-disciplinary approach for the assessment and treatment of misophonia. Treatment begins with a brief focus on the behavioral intervention, followed by the teaching of ACT skills to support the use of the behavioral methods. The intervention consists of 12 total individual sessions of ACT+behavioral management.
  Other Names: ACT
  Arms: Acceptance and commitment therapy
Behavioral: Progressive relaxation training — PRT for misophonia consists of basic psychoeducation for misophonia followed by PRT. PRT involves learning to tense and relax muscles. Early sessions focus on tensing and relaxing smaller muscle groups, while later sessions focus on larger muscle groups. Final sessions focus on relaxation as produced by recalling previous relaxation and a review of skills learned. PRT consists of 12 individual total sessions.
  Other Names: PRT
  Arms: Progressive relaxation training

SUMMARY:
The investigators are proposing to test Acceptance and Commitment Therapy (ACT)+ traditional audiological behavioral intervention as an integrated, multi-disciplinary approach for the assessment and treatment of misophonia. Participants will be 60 adults with misophonia and will be randomly assigned to receive 12 sessions of ACT+behavioral intervention or receive 12 weeks of progressive relaxation training+psychoeducation (PRT; a commonly used active control condition) after undergoing a comprehensive psychological and audiological evaluation.

DETAILED DESCRIPTION:
Acceptance and commitment therapy (ACT) is a promising psychotherapy for supporting traditional behavioral methods for treating misophonia, but has not been previously tested. ACT teaches skills to develop acceptance, mindfulness, and defusion from difficult internal experiences while increasing connections with personal values and encouraging meaningful behavioral changes.

This study will help determine if ACT+behavioral intervention is a feasible and acceptable treatment for misophonia, help clarify active psychological mechanisms of misophonia, and determine whether or not this combination of services can effectively help individuals diagnosed with misophonia.

ELIGIBILITY:
Inclusion Criteria:

* Individuals seeking treatment for misophonia.
* Meet clinical cut-off for misphonia (minimum score of five on the Misophonia Questionnaire).
* Stable on psychotropic medication for at least 30 days.
* English speaking.

Exclusion Criteria:

* Presence of psychological and/or neurological impairments that would preclude someone from participating in the study or exceed misophonia as the primary presenting problem (e.g. active self-harm or need for treatment for psychosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Misophonia Questionnaire | 9-12 months
  Self-report of misophonia symptoms. There are two subscales. The first subscale (misophonia symptoms) ranges from 0 to 76 and the second (misophonia severity) ranges from 1 to 15. For both subscales, higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Twohig, PhD, Principal Investigator — Utah State University
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: No